CLINICAL TRIAL: NCT00979615
Title: Safety and Efficacy of Olopatadine 0.6% and Azelastine 137 Mcg in Vasomotor Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Maria Tort, PhD, Manager, Global Medical Affairs, Alcon Research Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMA-09-03
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-04

CONDITIONS: Vasomotor Rhinitis
Keywords: vasomotor rhinitis; chronic non-allergic rhinitis; VMR
MeSH Terms: conditions — Rhinitis, Vasomotor | interventions — Olopatadine Hydrochloride; Nasal Sprays; azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Olopatadine HCL Nasal Spray, 0.6%
  Interventions: Drug: Olopatadine HCL (Patanase) Nasal Spray, 0.6%
- 2 (Active Comparator): Azelastine HCl Nasal Spray, 137 mcg
  Interventions: Drug: Azelastine HCl (Astelin) Nasal Spray, 137 mcg

INTERVENTIONS:
Drug: Olopatadine HCL (Patanase) Nasal Spray, 0.6% — 2 sprays/ nostril BID
  Arms: 1
Drug: Azelastine HCl (Astelin) Nasal Spray, 137 mcg — 2 sprays/ nostril BID
  Arms: 2

SUMMARY:
The purpose of this study is to examine safety and efficacy of Patanase and Astelin in treating the symptoms of non-allergic vasomotor rhinitis (VMR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of VMR with at least 2 years of chronic non-allergic rhinitis
* Negative skin tests to a panel of allergens and positive histamine test within last 2 years
* History of symptoms related to defined VMR triggers

Exclusion Criteria:

* Nasal disorder, surgery, or concurrent disease that could interfere with evaluation of study medications
* Bacterial or viral infection within 14 days of first visit. Diagnosis of acute sinusitis within 30 days of first visit
* Chronic use of drugs that can cause rhinitis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 9, 2009 - November 13, 2009
Groups:
- Olopatadine HCL: Olopatadine HCL Nasal Spray, 0.6%
- Azelastine HCl: Azelastine HCl Nasal Spray, 137 mcg
Period: Overall Study
Arm/Group | Olopatadine HCL | Azelastine HCl
Started | 63 | 66
Completed | 57 | 58
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olopatadine HCL | Azelastine HCl | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 51 | 54 | 105
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 85
  Male | 18 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in 2-week rTNSS From Baseline
Description: Change from baseline after 2 weeks in responses to patient-completed diaries for reflective Total Nasal VMR Symptom Scores (rTVSS). TVSS is composed of 4 individual assessments, which included nasal congestion, rhinorrhea, post nasal drip and sneezing; each of the 4 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 4 assessments are totaled for a composite score (TVSS score), the maximum of which could be 12. Reflective scores were assessed from the hour since the last dose of study medication.
Time Frame: 2 week
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCL | Azelastine HCl
Number analyzed (Participants) | 57 | 58
Units on a scale | 5.9 (3.0) | 6.5 (2.3)

2. Secondary Outcome: Mean Change in Rhinorrhea Reflective Score
Description: as for outcome 1
Time Frame: 2 week
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCL | Azelastine HCl
Number analyzed (Participants) | 44 | 43
Units on a scale | 1.5 (1.1) | 1.3 (1.0)

3. Secondary Outcome: Mean Change Postnasal Drip Reflective Score
Description: as for outcome 1
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCL | Azelastine HCl
Number analyzed (Participants) | 44 | 43
Units on a scale | 1.5 (1.2) | 1.8 (0.9)

4. Secondary Outcome: Mean Change Nasal Congestion Reflective Score
Description: as for outcome 1
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCL | Azelastine HCl
Number analyzed (Participants) | 44 | 43
Units on a scale | 1.4 (1.1) | 1.7 (1.2)

5. Secondary Outcome: Mean Change in Sneezing Reflective Score
Description: as for outcome 1
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCL | Azelastine HCl
Number analyzed (Participants) | 44 | 43
Units on a scale | 1.4 (0.9) | 1.7 (0.8)

ADVERSE EVENTS:
Time Frame: Two weeks
Arm/Group | Olopatadine HCL | Azelastine HCl
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/66
Other Adverse Events (participants affected / at risk) | 5/63 | 9/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olopatadine HCL (N=63) | Azelastine HCl (N=66)
Taste Disturbance (Gastrointestinal disorders) | 3 (3) | 6 (6)
Nose Bleeds (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No